CLINICAL TRIAL: NCT01789983
Title: Feasibility of an Evidence-based Walking Program in a Sample of Cancer Patients >60 Years of Age Undergoing Cytotoxic Chemotherapy
Brief Title: Feasibility of an Evidence-based Walking Program in Cancer Pts 60+ During Chemotherapy
Acronym: WWE
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1226; 12-1975 (Other: UNC IRB)
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Colon Cancer; Lung Cancer
Keywords: Physical Activity; Chemotherapy; Elderly; Geriatric; Walking; Geriatric Assessment; Geriatric Oncology
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms; Motor Activity | interventions — Walking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood Sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Breast Cancer Patients 60+: Breast Cancer Patients age 60 and older who have histologically confirmed stage I, II or III disease.
  Interventions: Behavioral: Walk With Ease Program; Other: Collect Blood, GA and Other Survey Tools
- Lung Cancer Patients 60+: Lung Cancer Patients age 60 and above who have stage I, II or III disease
  Interventions: Behavioral: Walk With Ease Program; Other: Collect Blood, GA and Other Survey Tools
- Colon Cancer Patients 60+: Colon cancer patients age 60 and above who have stage II or III disease.
  Interventions: Behavioral: Walk With Ease Program; Other: Collect Blood, GA and Other Survey Tools

INTERVENTIONS:
Behavioral: Walk With Ease Program — The primary activity required of study subjects is a 6-week self-directed (non-group) WWE walking program that study participants do at a place and time that is convenient for them. To start the intervention/program, we schedule a brief baseline meeting with study participants to discuss the program, provide the WWE workbook, secure printed informed consent, and complete various questionnaires. Study participants are also asked to maintain a daily walking diary that is provided to them.
  The WWE program includes a workbook with strengthening and stretching exercises, basic facts about arthritis and PA, and information on how to individualize the program.
  Other Names: WWE
Other: Collect Blood, GA and Other Survey Tools — * Geriatric Assessment (GA) (Version 5)
  * Functional Assessment of Cancer Therapy-General (FACT)
  * Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue36
  * Outcome Expectations for Exercise (OEE) scale29
  * Self-Efficacy to Manage Arthritis or Joint Pain (ASE/Arthritis Self-Efficacy)
  * Perceived Self-Efficacy for Fatigue Self-Management (PSEFSM)34,35
  * Visual Analog Scales (VAS)
  Surveys included in study are listed above. Whole Blood Sample will be collected for p16 analysis.

SUMMARY:
The study will look at conducting a medium-intense walking program called Walk With Ease with cancer patients age 60 and above who are starting chemotherapy treatment. We will measure how many of these patients complete their participation in this program.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the feasibility of implementing a moderate-intensity walking program (Walk With Ease/WWE) among cancer patients, age ≥60 years, as they undergo cytotoxic chemotherapy treatment. Feasibility will be determined based on the rate of participation in the WWE program. As secondary objectives, we will also establish the rate of completion of a number of instruments, including a Geriatric Assessment tool, and other instruments that measure self-reported quality of life (e.g., fatigue, depression, and pain), and self-reported physical activity (PA). Data from these instruments, as well as from serial measurements of a biomarker of aging (p16INK4a) will be explored and used to inform future studies designed to evaluate any relationship between these variables and participation in the WWE program.

We propose a sample (n=30) of cancer patients ≥60 years of age with potentially curable cancer and a diagnosis of Stage I-III breast cancer, Stage I-III lung cancer, or Stage II-III colon cancer, who are about to begin chemotherapy. Participation will be defined as completing the 6-week WWE program. Results from this study will be used in an RO1 application to the National Cancer Institute (NCI) pertaining to PA interventions among cancer patients and the effects of biomarkers on prognosis and survival.

ELIGIBILITY:
Inclusion Criteria:

* ≥60 years of age, male or female
* Histologically confirmed Stage I, II or III breast cancer (if the patient has had more than one breast cancer diagnosis, then the most recent diagnosis); Stage I, II or III lung cancer, or Stage II or III colon cancer
* Scheduled to begin a chemotherapy (or concomitant chemoradiotherapy) regimen that will last at least 6 weeks in duration
* English speaking
* IRB approved, signed written informed consent
* Approval from their treating physician to engage in moderate-intensity physical activity
* Patient-assessed ability to walk and engage in moderate physical activity
* Willing and able to meet all study requirements.

Exclusion Criteria:

* One or more significant medical conditions that in the physician's judgment preclude participation in the walking intervention
* Cancer surgery scheduled within the study period
* Unable to walk or engage in moderate-intensity physical activity

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colon, lung and breast cancer patients age 60 and above who are beginning chemotherapy or chemoradiation treatment.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
To measure the feasibility of implementing the WWE program among cancer patients, age ≥60, as they undergo cytotoxic chemotherapy treatment. | 1 year
  Feasibility will be defined as the proportion of recruited subjects who complete the 6-week WWE program.

SECONDARY OUTCOMES:
To measure the rate of completion of each of the following questionnaires/assessments at 3 different time points | 1 year
  The rate of completion of assessments will be measured at baseline, 6 weeks and end of chemotherapy treatment.
To measure relationships between physical activity levels and p16 levels. | 1 year
  To measure the association between number of minutes walked per day and number of times per week with p16 levels.

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Muss, MD, Principal Investigator — University of North Carolina Lineberger Comprehensive Cancer Center; Kirsten A Nyrop, PhD, Principal Investigator — University of North Carolina Thurston Arthritis Research Center
Locations (1):
- University of North Carolina Cancer Hospital, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: The Geriatric Oncology Research Program at UNC — https://unclineberger.org/patientcare/programs/geriatric